CLINICAL TRIAL: NCT02934373
Title: Evaluation of Subjective Ratings on a New Sound Processor and Compatible Products
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTD5665
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A New Sound Processor (Active Comparator): Sound Processor is the next generation sound processor.
  Interventions: Device: A New Sound Processor
- Subject's own sound processor (No Intervention)

INTERVENTIONS:
Device: A New Sound Processor
  Arms: A New Sound Processor

SUMMARY:
Clinical study designed to collect user feedback from Cochlear Implant recipients on a new Sound Processor System

ELIGIBILITY:
Inclusion Criteria:

1. 12 months old or older
2. Implanted with a CI24RE (Freedom implant) or later implant in at least one implanted ear
3. Use of the CP810, CP920 or CP910 sound processor
4. Willingness to participate in and to comply with all requirements of the protocol

Exclusion Criteria:

1. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks and limitations that are inherent to the procedure and prosthetic device
2. Additional disabilities or illnesses that would prevent participation in evaluations or compromise the integrity of the investigation or quality of data collected
3. Nucleus 22 or Nucleus 24 Implant in ear to be fitted with the investigational device

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Subjective rating with a new sound processor compared to ratings with each subjects own processor | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Brinson, Study Chair — Head of Clinical Affairs
Locations (3):
- SINT-Augustinus Antwerpen, Antwerp, Wilrijk, Belgium
- United Kingdom (2):
  - University of Southampton - Auditory Implant Service Highfield, Southampton, Hampshire
  - Nottingham University Hospitals - Queens Medical Centre, Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: No